CLINICAL TRIAL: NCT00318370
Title: A Study of the Efficacy of MORAb-003 in Subjects With Platinum-Sensitive Epithelial Ovarian Cancer in First Relapse
Brief Title: Effectiveness of MORAb-003 in Women With Ovarian Cancer Who Have Relapsed After Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-003-002
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Results first posted 2012-02-15 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Ovarian Cancer; Primary Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — farletuzumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Far Only (Experimental): Farletuzumab only (Far Only): farletuzumab, 100 milligrams (mg)/square meter (m2).
  Interventions: Drug: Farletuzumab
- Chemo Plus Far (Experimental): Chemo+Far: paclitaxel 175 mg/m2 (or docetaxel, 75 mg/m2) plus carboplatin area under the concentration-time curve (AUC) 5-6 intravenously (IV) on Day 1 of a 21-day cycle plus farletuzumab, 100 mg/m2.
  Interventions: Drug: Chemo Plus Far

INTERVENTIONS:
Drug: Farletuzumab — Weekly Farletuzumab infusions Dose dependent on dosing group
  Other Names: MORAb-003; Far Only
  Arms: Far Only
Drug: Chemo Plus Far — Chemo+Far: paclitaxel 175 mg/m2 (or docetaxel, 75 mg/m2) plus carboplatin area under the concentration-time curve (AUC) 5-6 intravenously (IV) on Day 1 of a 21-day cycle plus farletuzumab, 100 mg/m2.
  Arms: Chemo Plus Far

SUMMARY:
The purpose of this study is to determine if an investigational drug called MORAb-003 is useful by itself or when used with other approved cancer drugs in treating women with ovarian cancer. MORAb-003 is a monoclonal antibody directed against an antigen on most ovarian cancers.

DETAILED DESCRIPTION:
MORAb-003 is a monoclonal antibody that has the potential to be an effective agent against epithelial ovarian cancer (including primary fallopian tube and peritoneal adenocarcinoma) either alone or in combination with other drugs. MORAb-003 works by a different mechanism from other cancer therapeutics and has been shown to be well tolerated. This study allows the opportunity to determine if MORAb-003 can work either as a single agent

1. to treat a CA125-only relapse, or
2. in combination with standard platinum and taxane chemotherapy to treat a symptomatic relapse, and
3. to prolong a second response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects at least 18 years of age, with a histologically confirmed diagnosis of non-mucinous epithelial ovarian cancer (including fallopian tube and primary peritoneal cancer) in first relapse after a first remission of 6 to 18 months duration.
* Subjects must have undergone surgery. Subjects must have received primary chemotherapy, including at least one platinum agent.
* Subject is eligible for retreatment with the same chemotherapy regimen that was used to induce remission (Exception: may reduce the dose of or discontinue taxane if contraindicated due to neurotoxicity.)
* CA125 must have been elevated prior to original chemotherapy.
* CA125 must be elevated at the time of relapse.
* Life expectancy greater than or equal to 6 months, as estimated by the investigator.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2
* Subjects must consent to use a medically acceptable method of contraception throughout the study period and for 28 days after final MORAb-003 administration, unless surgically sterile.
* Any significant concomitant medical conditions must be well controlled and stable in the opinion of the investigator for at least 30 days prior to Study Day 1.
* Laboratory and clinical results within the 2 weeks prior to Study Day 1 as follows:

  * Absolute neutrophil count (ANC) ≥ 1.2 x 10e9/L
  * Platelet count ≥ 100 x 10e9/L
  * Hemoglobin ≥ 8 g/dL
* Subject must be willing and able to provide written informed consent. Translations of informed consent information may be provided, subject to the local institutional review board's (IRB's) policy.

Exclusion Criteria:

* Known central nervous system (CNS) tumor involvement.
* Evidence of other active malignancy requiring treatment.
* Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class III or IV, angina not well controlled by medication, or myocardial infarction within 6 months).
* Electrocardiogram (ECG) demonstrating clinically significant arrhythmias (Exception: Subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia [SVT], are eligible).
* Active serious systemic disease, including active bacterial or fungal infection.
* Active hepatitis or HIV infection.
* Treatment within three months with immunomodulatory therapy (e.g. interferons, immunoglobulin therapy, interleukin 1 receptor antagonist [IL-1RA] or systemic corticosteroids). Short term systemic corticosteroids or topical or intra-articular steroids are acceptable, subject to the judgment of the investigator.
* Treatment with a monoclonal antibody therapy AND have evidence of an immune or allergic reaction or documented HAHA.
* Maintenance of first remission by taxane or other chemotherapeutic agent(s).
* Initiation or planned initiation of cancer therapy not given to induce primary remission. Substitutions of agents materially similar to those used in the original regimen are permissible.
* Breast-feeding, pregnant, or likely to become pregnant during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-05; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan C. Weil, M.D., Study Director — Morphotek
Locations (20):
- United States (18):
  - Sharp HealthCare, San Diego, California
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Hematology and Oncology Specialists, LLC, Covington, Louisiana
  - Jayne Gurtler, M.D., Metairie, Louisiana
  - Hematology and Oncology Specialists, LLC, Metarie, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cooper University Hospital, Voorhees Township, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Lehigh Valley Women's Cancer Center, Allentown, Pennsylvania
  - Gynecology Oncology Research & Development, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - Peninsula Cancer Center, Newport News, Virginia
- Germany (2):
  - Krankenhaus Nordwest, Frankfurt
  - Nationales Centrum fur Tumorerkrankungen, Heidelberg

REFERENCES:
- [Derived] Armstrong DK, White AJ, Weil SC, Phillips M, Coleman RL. Farletuzumab (a monoclonal antibody against folate receptor alpha) in relapsed platinum-sensitive ovarian cancer. Gynecol Oncol. 2013 Jun;129(3):452-8. doi: 10.1016/j.ygyno.2013.03.002. Epub 2013 Mar 6. PMID 23474348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first 6 participants enrolled in this study were dosed at farletuzumab, 37.5 mg/m2. The next 6 participants were dosed at farletuzumab, 62.5 mg/m2. The remaining participants received farletuzumab, 100 mg/m2.
Groups:
- Chemo Plus Far: Platinum-based Chemotherapy plus farletuzumab (Chemo+Far): farletuzumab, 100 mg/m2 plus paclitaxel 175 mg/m2 (or docetaxel, 75 mg/m2) plus carboplatin area under the concentration-time curve (AUC) 5-6 intravenously (IV) on Day 1 of a 21-day cycle.
- Maintenance Far Only: Maintenance Far Only: farletuzumab, 100 milligrams (mg)/square meter (m2) for those subjects who completed Period 2, Chemo Plus Far.
Period: Period 1
Arm/Group | Far Only | Chemo Plus Far | Maintenance Far Only
Started | 28 | 0 | 0
Completed | 21 (21 participants proceeded from Far Only to Chemo Plus Far.) | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Period 2
Arm/Group | Far Only | Chemo Plus Far | Maintenance Far Only
Started | 0 | 47 (26 participants enrolled directly into Chemo Plus Far plus 21 participants from Far Only.) | 0
Completed | 0 | 36 | 0
Not Completed | 0 | 11 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 5 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Period: Period 3
Arm/Group | Far Only | Chemo Plus Far | Maintenance Far Only
Started | 0 | 0 | 36
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 33
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 24
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Other | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Far Only and Chemo Plus Far and Maintenance Far Only: Farletuzumab only (Far Only): farletuzumab, 100 milligrams (mg)/square meter (m2).
  Chemo+Far: paclitaxel 175 mg/m2 (or docetaxel, 75 mg/m2) plus carboplatin area under the concentration-time curve (AUC) 5-6 intravenously (IV) on Day 1 of a 21-day cycle plus farletuzumab, 100 mg/m2.
  Maintenance Far Only: farletuzumab, 100 milligrams (mg)/square meter (m2) for those subjects who completed the Period, Chemo Plus Far.
Arm/Group | Far Only and Chemo Plus Far and Maintenance Far Only
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
  Hispanic | 4

OUTCOME MEASURES:

1. Primary Outcome: Serologic Response (Change in CA125 Level)
Description: Defined using modified Gynecologic Cancer Intergroup (GCIG) criteria: Number of participants who achieved a 50% response = >50% decrease from baseline CA-125 (higher of 2 pretreatment CA-125 assessments and the level must be at least 52.5 kU/L).
Time Frame: Baseline to response (up to 30 weeks)
Population: All participants enrolled to initial farletuzumab only.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Far Only
Number analyzed (Participants) | 21
participants | 2 [0.9 to 23.5]

2. Primary Outcome: Serologic Response (Change in Cancer Antigen [CA-125] Level)
Description: Defined using modified Gynecologic Cancer Intergroup (GCIG) criteria: Number of participants who had a 50% response = >50% decrease from baseline CA-125 (higher of 2 pretreatment CA-125 assessments and the level must be at least 52.5 kU/L).
Time Frame: Baseline to response (up to 27 weeks)
Population: All participants enrolled to chemotherapy plus farletuzumab.
Measure: Number; unit: participants
Arm/Group | Chemo Plus Far
Number analyzed (Participants) | 47
participants | 41 [74.3 to 95.2]

3. Secondary Outcome: Time to Serologic Response (Change in CA-125 Level)
Description: Time to Serologic Response is defined as the time (weeks) from the date of first farletuzumab infusion to first documentation of 50% decrease from baseline CA-125 (higher of 2 pretreatment CA-125 assessments and at least twice the upper limit of normal) and then confirmed after 21 days.
Time Frame: Baseline to response (up to 27 weeks)
Population: All participants enrolled to intial chemotherapy plus farletuzumab.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chemo Plus Far
Number analyzed (Participants) | 47
Weeks | 3.3 [3.1 to 6.1]

4. Secondary Outcome: Duration of Serologic Response (CA-125)
Description: Calculated as the time from the first documentation of 50% or greater reduction in CA-125 to the first documentation of serologic progression or death due to any cause. Serologic progression was defined as the first date of the CA-125 level being >2 X ULN on two occasions.
Time Frame: Baseline to response (up to 44 months)
Population: All participants enrolled to initial chemotherapy plus farletuzumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemo Plus Far
Number analyzed (Participants) | 47
Months | NA [9.9 to NA] — NA = Not Estimable because the median number of participants did not progress or die.

5. Secondary Outcome: Overall Response Rate
Description: The Overall Response Rate (ORR) will be determined by applying standard RECIST criteria to objective measures of disease, such as CT or MRI scans. Participants will be assigned to one of the categories of change in disease status, namely, "complete response" (CR), "partial response" (PR), "stable disease" (SD), or "progressive disease" (PD). ORR is defined as the percentage of participants with objective evidence of CR or PR.
Time Frame: Baseline to response (up to 44 months)
Measure: Number; unit: percentage of participants
Arm/Group | Chemo Plus Far
Number analyzed (Participants) | 47
percentage of participants
  Complete Response | 6.8
  Partial Response | 63.6
  Stable Disease | 20.5
  Progressive Disease | 4.5
  Not Evaluable | 6.8

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined for participants treated in Chemo Plus Far as the time (in months) from date of first dose in Chemo Plus Far until date of the first observation of progression based on first date of the CA-125 >2 X ULN on two occasions, or date of death, whatever the cause. If progression or death is not observed for a participant, the PFS time is censored at the later date of last tumor assessment or CA125 assessment without evidence of progression prior to the date of initiation of further anti-tumor treatment.
Time Frame: Baseline to response (up to 44 months)
Population: All participants who received chemotherapy plus farletuzumab as well as those who continued on maintenance farletuzumab.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Chemo Plus Far Plus Maintenance Far Only: Platinum-based Chemotherapy plus farletuzumab (Chemo+Far): farletuzumab, 100 mg/m2 plus paclitaxel 175 mg/m2 (or docetaxel, 75 mg/m2) plus carboplatin area under the concentration-time curve (AUC) 5-6 intravenously (IV) on Day 1 of a 21-day cycle.
  Maintenace Far Only: farletuzumab, 100 mg/m2
Arm/Group | Chemo Plus Far Plus Maintenance Far Only
Number analyzed (Participants) | 47
Months | 10.2 [7.4 to 13.1]

7. Secondary Outcome: Percentage of Participants Who Had a Prolongation of Remission
Description: Percentage of participants whose second remission was longer than their first remission. The length of remission will be determined for participants who attain CR or PR (or SD and investigator's assessment of clinical benefit). Prolongation of remission will be defined as a length of remission occurring on this study that is ≥ 1 day longer than the length of remission to the original therapy. The length of remission on this study (second remission) will be defined as the amount of time from the date of first CR or PR to the end of this remission.
Time Frame: Baseline to response (up to 44 months)
Population: All participants who received chemotherapy plus farletuzumab as well as those who continued on maintenance farletuzumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemo Plus Far Plus Maintenance Far Only
Number analyzed (Participants) | 39
percentage of participants | 25.6 [13.0 to 42.1]

ADVERSE EVENTS:
Arm/Group | Far Only and Chemo Plus Far and Maintenance Far Only
Serious Adverse Events (participants affected / at risk) | 20/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Far Only and Chemo Plus Far and Maintenance Far Only (N=54)
Abdominal Pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Large intestinal obstruction (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Rectal haemorrohage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Urosepsis (Infections and infestations) | 2
Clostridium colitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Adverse drug reaction (General disorders) | 1
Chest discomfort (General disorders) | 1
Injection site reaction (General disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Peripheral occlusive disease (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Psychiatric evaluation (Investigations) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydronephrosis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Far Only and Chemo Plus Far and Maintenance Far Only (N=54)
Nausea (Gastrointestinal disorders) | 35
Constipation (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 25
Abdominal Pain (Gastrointestinal disorders) | 24
Abdominal distension (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 4
Hiatus hernia (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 3
Abdominal tenderness (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 51
Pyrexia (General disorders) | 22
Chills (General disorders) | 14
Oedema peripheral (General disorders) | 14
Asthenia (General disorders) | 9
Adverse drug reaction (General disorders) | 8
Pain (General disorders) | 7
Chest discomfort (General disorders) | 5
Influenza-like illness (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Chest pain (General disorders) | 3
Infusion site pain (General disorders) | 3
Malaise (General disorders) | 3
Urinary tract infection (Infections and infestations) | 19
Nasopharyngitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Headache (Nervous system disorders) | 27
Dizziness (Nervous system disorders) | 11
Neuropathy peripheral (Nervous system disorders) | 8
Neuropathy (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 23
Neutropenia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 3
Red blood cell count decreased (Investigations) | 3
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 8
Hypertension (Vascular disorders) | 6
Flushing (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4
Hot flush (Vascular disorders) | 3
Haematuria (Renal and urinary disorders) | 8
Dysuria (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 5
Tachycardia (Cardiac disorders) | 3
Lacrimation increased (Eye disorders) | 4
Vision blurred (Eye disorders) | 4
Ear pain (Ear and labyrinth disorders) | 5
Vertigo (Ear and labyrinth disorders) | 5
Seasonal allergy (Immune system disorders) | 4
Cytokine release syndrome (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less